CLINICAL TRIAL: NCT06723197
Title: Efficacy of Different Durations of Dual and Quadruple Regimens for Helicobacter Pylori Eradication: a Multicentre, Randomised, Controlled Trial
Brief Title: Efficacy of Different Durations of Dual and Quadruple Regimens for Helicobacter Pylori Eradication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Zibo Maternal and Child Health Hospital (Unknown); Zaozhuang Municipal Hospital (Other); Feicheng Municipal People's Hospital (Unknown); Shandong University of Traditional Chinese Medicine (Other); The People's Hospital of Jimo.Qingdao (Unknown); Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Ph.D, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202411
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: HELICOBACTER PYLORI INFECTIONS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 14-day dual regimen (Active Comparator)
  Interventions: Drug: vonoprazan+amoxicillin; Other: Duration of eradication regimen: 14-day
- 10-day dual regimen (Experimental)
  Interventions: Drug: vonoprazan+amoxicillin; Other: Duration of eradication regimen: 10-day
- 7-day quadruple regimen (Experimental)
  Interventions: Other: Duration of eradication regimen: 7-day; Drug: vonoprazan+amoxicillin+tetracycline+bismuth

INTERVENTIONS:
Drug: vonoprazan+amoxicillin — Drug combinations for dual regimens：vonoprazan+amoxicillin
  Arms: 10-day dual regimen; 14-day dual regimen
Other: Duration of eradication regimen: 7-day — Duration of eradication regimen: 7-day
  Arms: 7-day quadruple regimen
Drug: vonoprazan+amoxicillin+tetracycline+bismuth — Drug combinations for quadruple regimens: vonoprazan+amoxicillin+tetracycline+bismuth
  Arms: 7-day quadruple regimen
Other: Duration of eradication regimen: 10-day — Duration of eradication regimen: 10-day
  Arms: 10-day dual regimen
Other: Duration of eradication regimen: 14-day — Duration of eradication regimen: 14-day
  Arms: 14-day dual regimen

SUMMARY:
The study aimed to compare the efficacy and safety of dual and quadruple regimens with different durations (7-day, 10-day, 14-day) for the eradication of Helicobacter pylori. Subjects were randomized to receive the intervention and were reviewed by 13C-urea breath test after 6 weeks. The eradication rates, adverse reaction rates and patient adherence were calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years old
2. Patients with H.pylori infection (13C/14C-urea breath test)
3. Patients without previous treatment for H. pylori eradication

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%
2. Patients with active gastrointestinal bleeding
3. Patients with a history of upper gastrointestinal surgery
4. Patients allergic to treatment drugs
5. Patients with medication history of bismuth, antibiotics within 4 weeks, or proton pump inhibitor within 2 weeks
6. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
8. Patients who are unwilling or incapable to provide informed consents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Six weeks after treatment
  13C-urea breath test was used to determine whether eradication was successful. Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in the three groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after treatment
  Drug-related adverse reactions needs to be recorded after treatment
Patient compliance | Immediately after treatment
  The number of missed and overdosed doses of medication needs to be completed after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qian HS, Li WJ, Dang YN, Li LR, Xu XB, Yuan L, Zhang WF, Yang Z, Gao X, Zhang M, Li X, Zhang GX. Ten-Day Vonoprazan-Amoxicillin Dual Therapy as a First-Line Treatment of Helicobacter pylori Infection Compared With Bismuth-Containing Quadruple Therapy. Am J Gastroenterol. 2023 Apr 1;118(4):627-634. doi: 10.14309/ajg.0000000000002086. Epub 2022 Dec 2. PMID 36729890
- [Background] Du RC, Hu YX, Ouyang Y, Ling LX, Xu JY, Sa R, Liu XS, Hong JB, Zhu Y, Lu NH, Hu Y. Vonoprazan and amoxicillin dual therapy as the first-line treatment of Helicobacter pylori infection: A systematic review and meta-analysis. Helicobacter. 2024 Jan-Feb;29(1):e13039. doi: 10.1111/hel.13039. Epub 2023 Nov 30. PMID 38036941
- [Background] Zhou L, Lu H, Song Z, Lyu B, Chen Y, Wang J, Xia J, Zhao Z; on behalf of Helicobacter Pylori Study Group of Chinese Society of Gastroenterology. 2022 Chinese national clinical practice guideline on Helicobacter pylori eradication treatment. Chin Med J (Engl). 2022 Dec 20;135(24):2899-2910. doi: 10.1097/CM9.0000000000002546. PMID 36579940
- [Background] Crowe SE. Helicobacter pylori Infection. N Engl J Med. 2019 Mar 21;380(12):1158-1165. doi: 10.1056/NEJMcp1710945. No abstract available. PMID 30893536
- [Background] Li Y, Choi H, Leung K, Jiang F, Graham DY, Leung WK. Global prevalence of Helicobacter pylori infection between 1980 and 2022: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2023 Jun;8(6):553-564. doi: 10.1016/S2468-1253(23)00070-5. Epub 2023 Apr 20. PMID 37086739